CLINICAL TRIAL: NCT03137303
Title: Reducing Diagnostic Error to Improve Patient Safety in COPD and Asthma (REDEFINE Study)
Acronym: REDEFINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Min Joo, MD MPH, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-1209
Record Dates: First submitted 2017-04-14; First posted 2017-05-02 (Actual); Results first posted 2021-07-22 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: COPD Asthma
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Subject Usual Care (Placebo Comparator): On the day of the outpatient visit, subjects will be advised to arrive 90 minutes prior to their clinic visit. The following will be performed.
  1. Subject demographic and contact information
  2. Co-morbid conditions
  3. Smoking history
  4. Medication history from patient and also from pharmacy used by subjects
  5. A respiratory exacerbation history in the past year
  6. Modified Medical Research Counsel (mMRC) dyspnea scale
  7. Quality of life measures
  Subjects will be advised to go to their clinics and be managed by their PCP thereafter.
  At the end of the 1 year followup, the patient will be scheduled for a pre and post BD spirometry and undergo the same spirometry protocol as the intervention group.
  Interventions: Drug: Albuterol; Device: Spirometry at 12-month follow-up
- Patient-Subject Intervention (Experimental): On the day of the outpatient visit, subjects will be advised to arrive 90 minutes prior to their clinic visit in the same building as the clinic site. The following information will be collected and procedures will be performed:
  1. Subject demographic and contact information
  2. Co-morbid conditions
  3. Smoking history
  4. Medication history from patient and also from pharmacy used by subjects
  5. A respiratory exacerbation history in the past year
  6. Modified Medical Research Counsel (mMRC) dyspnea scale
  7. Quality of life measures
  8. Pre and post-bronchodilator using Albuterol (BD) spirometry
  Interventions: Device: Spirometry at initial visit; Drug: Albuterol

INTERVENTIONS:
Device: Spirometry at initial visit — Initial visit for the intervention group, an initial demographics form and health questionnaires. To evaluate the breathing, a pre and post broncho dilator will be performed as well as a spirometry test.
  Other Names: KoKo Spirometer (Model 313120); 3 Liter Calibration Syringe
  Arms: Patient-Subject Intervention
Drug: Albuterol — The post broncho dilator spirometry test will be preformed after a breathing medication called Albuterol. Albuterol is used in standard practice for COPD and is commonly used during spirometry.
  Other Names: Albuterol, Ventolin, Proventil, Accuneb
Device: Spirometry at 12-month follow-up — At the end of the 1 year followup, the patient will be scheduled for a pre and post BD spirometry test and undergo the same spirometry protocol as the intervention group.
  Other Names: KoKo Spirometer (Model 313120); 3 Liter Calibration Syringe
  Arms: Patient Subject Usual Care

SUMMARY:
The purpose of this study is to evaluate the use of spirometry in identifying Diagnostic Error in COPD and Asthma patients.

DETAILED DESCRIPTION:
Asthma and chronic obstructive pulmonary disease (COPD) are common chronic lung diseases that are diagnosed in more than 30 million adults in the United States. However, diagnostic error (DE), is considered one of the most common and harmful of patient-safety problems by the Institute of Medicine, occur frequently with asthma and/or COPD and disproportionately affect minorities and the under-served. DE leads to lost opportunities to identify other chronic conditions, avoidable morbidity and mortality, unnecessary costs to patients and health systems, and poor quality of care. Shortness of breath or dyspnea, which is a common symptom in asthma and COPD, is also common for many other chronic conditions such as cardiovascular disease and obesity. A better understanding of the impact of DE and interventions to improve diagnostic accuracy in asthma and COPD are of particular importance for minorities and the under-served that are disproportionately affected by conditions leading to dyspnea.

Spirometry is a simple, mobile, and essential test that is recommended by all major national and international guidelines for the diagnosis of asthma and COPD. However it is well known that spirometry is not routinely used in the ambulatory primary care setting and minorities and the underserved population are less likely to have spirometry leading to greater prevalence of DE. It has been estimated that 30-50% of people with an existing diagnosis of asthma and COPD were found to be misdiagnosed. Many of these patients misdiagnosed with asthma and/or COPD receive unnecessary respiratory pharmacotherapy which can pose serious risks including pneumonia, cardiovascular events, and mortality. In the setting of DE, these are considered avoidable and unnecessary respiratory pharmacotherapy use in minorities and the underserved that are already disproportionately affected by cardiovascular disease increases the risk of poorer outcomes. There is also DE in the diagnosis of asthma versus COPD, as these are both clinically distinct respiratory disorders with nuances in treatment recommendations. It is reported that African-Americans are considered to have increasing COPD mortality and are disproportionately affected by asthma death rates. However, as spirometry is not routinely performed and DE is prevalent in asthma and COPD, a component of these poor outcomes may be attributable to missed or delayed diagnoses of other chronic conditions or misdiagnosis within asthma and COPD.

Barriers to the use of spirometry in primary care exist at provider and health systems levels. Previous studies show that primary care providers (PCPs) lack knowledge in existing guidelines and in implementing spirometry into primary care clinics. Beyond these barriers, PCPs struggle with logistical challenges such as time and workflow constraints with clinic visits lasting 15 minutes or less in patients with multiple chronic medical conditions. These predisposing and enabling factors explain why prior studies that included interventions to educate PCPs and incorporate spirometry by training personnel in primary care clinics have had limited results.

A new paradigm to improve guideline based care for asthma and COPD which includes spirometry is needed and can lead to a better understanding of DE and improved patient safety and patient-centered outcomes. Health Promoters or Community health workers (CHWs) have been supplementing medical care by disseminating appropriate health care practices for underserved minority populations. However, studies which include diagnostic evaluations with spirometry for asthma and COPD have not been performed. The REDEFINE program (Reducing Diagnostic Error to Improve PatieNt SafEty in COPD and Asthma) will incorporate health promoters working collaboratively with PCPs to address identified barriers to guideline based care which includes spirometry for the diagnosis of asthma and COPD for patients at risk for DE. We propose a comparative effectiveness study to better understand the epidemiology of DE and to evaluate the effectiveness and economic impact of providing the REDEFINE program to an underserved, predominantly minority population with a diagnosis of asthma and/or COPD at risk for DE.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥40 years of age
* 2. Use of a maintenance respiratory medication and one of the following in the past year:
* 3. Diagnosis of asthma and/or COPD
* 4. No spirometry test performed in the past 3 years
* 5. Past or current smoker or is exposed to tobacco

Exclusion Criteria:

* Unable to perform adequate spirometry
* Non-English speaking
* Pregnancy
* Plans to move from the Chicago Area within the next year
* Seen by pulmonary specialist in the past 3 years
* Any terminal illness with a life expectancy of <6 months
* Life threatening (e.g. intensive care admission and/or use of mechanical ventilation) respiratory failure event in the past year.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min Joo, MD MPH, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - CCHHS, Chicago, Illinois
  - UI Health, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Center for Health Statistics. Chronic Obstructive Pulmonary Disease Among Adults Aged 18 and Over in the United States, 1998-2009. 2011
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: asthma prevalence, disease characteristics, and self-management education: United States, 2001--2009. MMWR Morb Mortal Wkly Rep. 2011 May 6;60(17):547-52. PMID 21544044
- [Background] Ball JR, Balogh E. Improving Diagnosis in Health Care: Highlights of a Report From the National Academies of Sciences, Engineering, and Medicine. Ann Intern Med. 2016 Jan 5;164(1):59-61. doi: 10.7326/M15-2256. Epub 2015 Sep 29. No abstract available. PMID 26414299
- [Background] Committee on Diagnostic Error in Health Care; Board on Health Care Services; Institute of Medicine; The National Academies of Sciences, Engineering, and Medicine; Balogh EP, Miller BT, Ball JR, editors. Improving Diagnosis in Health Care. Washington (DC): National Academies Press (US); 2015 Dec 29. Available from http://www.ncbi.nlm.nih.gov/books/NBK338596/ PMID 26803862
- [Background] Singh H, Graber ML. Improving Diagnosis in Health Care--The Next Imperative for Patient Safety. N Engl J Med. 2015 Dec 24;373(26):2493-5. doi: 10.1056/NEJMp1512241. Epub 2015 Nov 11. No abstract available. PMID 26559457
- [Background] Khullar D, Jha AK, Jena AB. Reducing Diagnostic Errors--Why Now? N Engl J Med. 2015 Dec 24;373(26):2491-3. doi: 10.1056/NEJMp1508044. Epub 2015 Sep 23. No abstract available. PMID 26397948
- [Background] Global Initiative for Asthma. Global strategy for asthma management and prevention. Bethesda, MD, USA: GINA;2015
- [Background] Qaseem A, Wilt TJ, Weinberger SE, Hanania NA, Criner G, van der Molen T, Marciniuk DD, Denberg T, Schunemann H, Wedzicha W, MacDonald R, Shekelle P; American College of Physicians; American College of Chest Physicians; American Thoracic Society; European Respiratory Society. Diagnosis and management of stable chronic obstructive pulmonary disease: a clinical practice guideline update from the American College of Physicians, American College of Chest Physicians, American Thoracic Society, and European Respiratory Society. Ann Intern Med. 2011 Aug 2;155(3):179-91. doi: 10.7326/0003-4819-155-3-201108020-00008. PMID 21810710
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Bolton CE, Ionescu AA, Edwards PH, Faulkner TA, Edwards SM, Shale DJ. Attaining a correct diagnosis of COPD in general practice. Respir Med. 2005 Apr;99(4):493-500. doi: 10.1016/j.rmed.2004.09.015. Epub 2004 Nov 11. PMID 15763457
- [Background] Damarla M, Celli BR, Mullerova HX, Pinto-Plata VM. Discrepancy in the use of confirmatory tests in patients hospitalized with the diagnosis of chronic obstructive pulmonary disease or congestive heart failure. Respir Care. 2006 Oct;51(10):1120-4. PMID 17005056
- [Background] Han MK, Kim MG, Mardon R, Renner P, Sullivan S, Diette GB, Martinez FJ. Spirometry utilization for COPD: how do we measure up? Chest. 2007 Aug;132(2):403-9. doi: 10.1378/chest.06-2846. Epub 2007 Jun 5. PMID 17550936
- [Background] Lee TA, Bartle B, Weiss KB. Spirometry use in clinical practice following diagnosis of COPD. Chest. 2006 Jun;129(6):1509-15. doi: 10.1378/chest.129.6.1509. PMID 16778268
- [Background] Mapel DW, Picchi MA, Hurley JS, Frost FJ, Petersen HV, Mapel VM, Coultas DB. Utilization in COPD: patient characteristics and diagnostic evaluation. Chest. 2000 May;117(5 Suppl 2):346S-53S. doi: 10.1378/chest.117.5_suppl_2.346s. PMID 10843975
- [Background] Miravitlles M, de la Roza C, Naberan K, Lamban M, Gobartt E, Martin A. Use of spirometry and patterns of prescribing in COPD in primary care. Respir Med. 2007 Aug;101(8):1753-60. doi: 10.1016/j.rmed.2007.02.019. Epub 2007 Apr 19. PMID 17448651
- [Background] Mularski RA, Asch SM, Shrank WH, Kerr EA, Setodji CM, Adams JL, Keesey J, McGlynn EA. The quality of obstructive lung disease care for adults in the United States as measured by adherence to recommended processes. Chest. 2006 Dec;130(6):1844-50. doi: 10.1378/chest.130.6.1844. PMID 17167007
- [Background] Walters JA, Hansen E, Mudge P, Johns DP, Walters EH, Wood-Baker R. Barriers to the use of spirometry in general practice. Aust Fam Physician. 2005 Mar;34(3):201-3. PMID 15799676
- [Background] O'Dowd LC, Fife D, Tenhave T, Panettieri RA Jr. Attitudes of physicians toward objective measures of airway function in asthma. Am J Med. 2003 Apr 1;114(5):391-6. doi: 10.1016/s0002-9343(03)00007-x. PMID 12714129
- [Background] Ghattas C, Dai A, Gemmel DJ, Awad MH. Over diagnosis of chronic obstructive pulmonary disease in an underserved patient population. Int J Chron Obstruct Pulmon Dis. 2013;8:545-9. doi: 10.2147/COPD.S45693. Epub 2013 Nov 12. PMID 24348030
- [Background] Prieto-Centurion V, Rolle AJ, Au DH, Carson SS, Henderson AG, Lee TA, Lindenauer PK, McBurnie MA, Mularski RA, Naureckas ET, Vollmer WM, Joese BJ, Krishnan JA; CONCERT Consortium. Multicenter study comparing case definitions used to identify patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2014 Nov 1;190(9):989-95. doi: 10.1164/rccm.201406-1166OC. PMID 25192554
- [Background] Han MK, Postma D, Mannino DM, Giardino ND, Buist S, Curtis JL, Martinez FJ. Gender and chronic obstructive pulmonary disease: why it matters. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1179-84. doi: 10.1164/rccm.200704-553CC. Epub 2007 Aug 2. PMID 17673696
- [Background] Chapman KR, Tashkin DP, Pye DJ. Gender bias in the diagnosis of COPD. Chest. 2001 Jun;119(6):1691-5. doi: 10.1378/chest.119.6.1691. PMID 11399692
- [Background] Franks P, Clancy CM, Naumburg EH. Sex, access, and excess. Ann Intern Med. 1995 Oct 1;123(7):548-50. doi: 10.7326/0003-4819-123-7-199510010-00012. No abstract available. PMID 7661501
- [Background] Ohar J, Fromer L, Donohue JF. Reconsidering sex-based stereotypes of COPD. Prim Care Respir J. 2011 Dec;20(4):370-8. doi: 10.4104/pcrj.2011.00070. PMID 21922124
- [Background] Tinkelman DG, Price DB, Nordyke RJ, Halbert RJ. Misdiagnosis of COPD and asthma in primary care patients 40 years of age and over. J Asthma. 2006 Jan-Feb;43(1):75-80. doi: 10.1080/02770900500448738. PMID 16448970
- [Background] Abramson MJ, Schattner RL, Sulaiman ND, Del Colle EA, Aroni R, Thien F. Accuracy of asthma and COPD diagnosis in Australian general practice: a mixed methods study. Prim Care Respir J. 2012 Jun;21(2):167-73. doi: 10.4104/pcrj.2011.00103. PMID 22234387
- [Background] Melbye H, Drivenes E, Dalbak LG, Leinan T, Hoegh-Henrichsen S, Ostrem A. Asthma, chronic obstructive pulmonary disease, or both? Diagnostic labeling and spirometry in primary care patients aged 40 years or more. Int J Chron Obstruct Pulmon Dis. 2011;6:597-603. doi: 10.2147/COPD.S25955. Epub 2011 Nov 17. PMID 22135492
- [Background] Griffiths C, Feder G, Wedzicha J, Foster G, Livingstone A, Marlowe GS. Feasibility of spirometry and reversibility testing for the identification of patients with chronic obstructive pulmonary disease on asthma registers in general practice. Respir Med. 1999 Dec;93(12):903-8. doi: 10.1016/s0954-6111(99)90057-4. PMID 10653053
- [Background] Sichletidis L, Chloros D, Spyratos D, Chatzidimitriou N, Chatziiliadis P, Protopappas N, Charalambidou O, Pelagidou D, Zarvalis E, Patakas D. The validity of the diagnosis of chronic obstructive pulmonary disease in general practice. Prim Care Respir J. 2007 Apr;16(2):82-8. doi: 10.3132/pcrj.2007.00016. PMID 17377688
- [Background] Walters JA, Walters EH, Nelson M, Robinson A, Scott J, Turner P, Wood-Baker R. Factors associated with misdiagnosis of COPD in primary care. Prim Care Respir J. 2011 Dec;20(4):396-402. doi: 10.4104/pcrj.2011.00039. PMID 21687918
- [Background] Buffels J, Degryse J, Liistro G, Decramer M. Differential diagnosis in a primary care population with presumed airway obstruction: a real-life study. Respiration. 2012;84(1):44-54. doi: 10.1159/000332836. Epub 2011 Nov 15. PMID 22094827
- [Background] Nelson HS, Weiss ST, Bleecker ER, Yancey SW, Dorinsky PM; SMART Study Group. The Salmeterol Multicenter Asthma Research Trial: a comparison of usual pharmacotherapy for asthma or usual pharmacotherapy plus salmeterol. Chest. 2006 Jan;129(1):15-26. doi: 10.1378/chest.129.1.15. PMID 16424409
- [Background] Lee TA, Pickard AS, Au DH, Bartle B, Weiss KB. Risk for death associated with medications for recently diagnosed chronic obstructive pulmonary disease. Ann Intern Med. 2008 Sep 16;149(6):380-90. doi: 10.7326/0003-4819-149-6-200809160-00004. PMID 18794557
- [Background] Singh S, Loke YK, Furberg CD. Inhaled anticholinergics and risk of major adverse cardiovascular events in patients with chronic obstructive pulmonary disease: a systematic review and meta-analysis. JAMA. 2008 Sep 24;300(12):1439-50. doi: 10.1001/jama.300.12.1439. PMID 18812535
- [Background] Van den Bruel A, Gailly J, Neyt M. Does tiotropium lower exacerbation and hospitalization frequency in COPD patients: results of a meta-analysis. BMC Pulm Med. 2010 Sep 21;10:50. doi: 10.1186/1471-2466-10-50. PMID 20858226
- [Background] Ogale SS, Lee TA, Au DH, Boudreau DM, Sullivan SD. Cardiovascular events associated with ipratropium bromide in COPD. Chest. 2010 Jan;137(1):13-9. doi: 10.1378/chest.08-2367. Epub 2009 Apr 10. PMID 19363211
- [Background] Macie C, Wooldrage K, Manfreda J, Anthonisen N. Cardiovascular morbidity and the use of inhaled bronchodilators. Int J Chron Obstruct Pulmon Dis. 2008;3(1):163-9. doi: 10.2147/copd.s1516. PMID 18488440
- [Background] Ringbaek T, Viskum K. Is there any association between inhaled ipratropium and mortality in patients with COPD and asthma? Respir Med. 2003 Mar;97(3):264-72. doi: 10.1053/rmed.2003.1423. PMID 12645834
- [Background] Guite HF, Dundas R, Burney PG. Risk factors for death from asthma, chronic obstructive pulmonary disease, and cardiovascular disease after a hospital admission for asthma. Thorax. 1999 Apr;54(4):301-7. doi: 10.1136/thx.54.4.301. PMID 10092690
- [Background] Singh S, Loke YK, Enright PL, Furberg CD. Mortality associated with tiotropium mist inhaler in patients with chronic obstructive pulmonary disease: systematic review and meta-analysis of randomised controlled trials. BMJ. 2011 Jun 14;342:d3215. doi: 10.1136/bmj.d3215. PMID 21672999
- [Background] Martin-Merino E, Garcia-Rodriguez LA, Masso-Gonzalez EL, Roehrborn CG. Do oral antimuscarinic drugs carry an increased risk of acute urinary retention? J Urol. 2009 Oct;182(4):1442-8. doi: 10.1016/j.juro.2009.06.051. Epub 2009 Aug 15. PMID 19683302
- [Background] Armitage JN, Sibanda N, Cathcart PJ, Emberton M, van der Meulen JH. Mortality in men admitted to hospital with acute urinary retention: database analysis. BMJ. 2007 Dec 8;335(7631):1199-202. doi: 10.1136/bmj.39377.617269.55. Epub 2007 Nov 8. PMID 17991937
- [Background] Calverley PM, Anderson JA, Celli B, Ferguson GT, Jenkins C, Jones PW, Yates JC, Vestbo J; TORCH investigators. Salmeterol and fluticasone propionate and survival in chronic obstructive pulmonary disease. N Engl J Med. 2007 Feb 22;356(8):775-89. doi: 10.1056/NEJMoa063070. PMID 17314337
- [Background] Ernst P, Gonzalez AV, Brassard P, Suissa S. Inhaled corticosteroid use in chronic obstructive pulmonary disease and the risk of hospitalization for pneumonia. Am J Respir Crit Care Med. 2007 Jul 15;176(2):162-6. doi: 10.1164/rccm.200611-1630OC. Epub 2007 Mar 30. PMID 17400730
- [Background] Kardos P, Wencker M, Glaab T, Vogelmeier C. Impact of salmeterol/fluticasone propionate versus salmeterol on exacerbations in severe chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2007 Jan 15;175(2):144-9. doi: 10.1164/rccm.200602-244OC. Epub 2006 Oct 19. PMID 17053207
- [Background] Ferguson GT, Anzueto A, Fei R, Emmett A, Knobil K, Kalberg C. Effect of fluticasone propionate/salmeterol (250/50 microg) or salmeterol (50 microg) on COPD exacerbations. Respir Med. 2008 Aug;102(8):1099-108. doi: 10.1016/j.rmed.2008.04.019. Epub 2008 Jul 9. PMID 18614347
- [Background] Wedzicha JA, Calverley PM, Seemungal TA, Hagan G, Ansari Z, Stockley RA; INSPIRE Investigators. The prevention of chronic obstructive pulmonary disease exacerbations by salmeterol/fluticasone propionate or tiotropium bromide. Am J Respir Crit Care Med. 2008 Jan 1;177(1):19-26. doi: 10.1164/rccm.200707-973OC. Epub 2007 Oct 4. PMID 17916806
- [Background] Joo MJ, Au DH, Fitzgibbon ML, Lee TA. Inhaled corticosteroids and risk of pneumonia in newly diagnosed COPD. Respir Med. 2010 Feb;104(2):246-52. doi: 10.1016/j.rmed.2009.10.002. Epub 2009 Oct 30. PMID 19879745
- [Background] Yawn BP, Li Y, Tian H, Zhang J, Arcona S, Kahler KH. Inhaled corticosteroid use in patients with chronic obstructive pulmonary disease and the risk of pneumonia: a retrospective claims data analysis. Int J Chron Obstruct Pulmon Dis. 2013;8:295-304. doi: 10.2147/COPD.S42366. Epub 2013 Jun 27. PMID 23836970
- [Background] McKeever T, Harrison TW, Hubbard R, Shaw D. Inhaled corticosteroids and the risk of pneumonia in people with asthma: a case-control study. Chest. 2013 Dec;144(6):1788-1794. doi: 10.1378/chest.13-0871. PMID 23990003
- [Background] Lee TA, Weiss KB. Fracture risk associated with inhaled corticosteroid use in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Apr 1;169(7):855-9. doi: 10.1164/rccm.200307-926OC. Epub 2004 Jan 7. PMID 14711795
- [Background] Mensah GA, Mokdad AH, Ford ES, Greenlund KJ, Croft JB. State of disparities in cardiovascular health in the United States. Circulation. 2005 Mar 15;111(10):1233-41. doi: 10.1161/01.CIR.0000158136.76824.04. PMID 15769763
- [Background] Cooper R, Cutler J, Desvigne-Nickens P, Fortmann SP, Friedman L, Havlik R, Hogelin G, Marler J, McGovern P, Morosco G, Mosca L, Pearson T, Stamler J, Stryer D, Thom T. Trends and disparities in coronary heart disease, stroke, and other cardiovascular diseases in the United States: findings of the national conference on cardiovascular disease prevention. Circulation. 2000 Dec 19;102(25):3137-47. doi: 10.1161/01.cir.102.25.3137. PMID 11120707
- [Background] Ski CF, King-Shier KM, Thompson DR. Gender, socioeconomic and ethnic/racial disparities in cardiovascular disease: a time for change. Int J Cardiol. 2014 Jan 1;170(3):255-7. doi: 10.1016/j.ijcard.2013.10.082. Epub 2013 Nov 1. PMID 24238906
- [Background] Akinbami LJ, Moorman JE, Bailey C, Zahran HS, King M, Johnson CA, Liu X. Trends in asthma prevalence, health care use, and mortality in the United States, 2001-2010. NCHS Data Brief. 2012 May;(94):1-8. PMID 22617340
- [Background] Morbidity & Mortality: 2012 Chart Book on Cardiovascular, Lung, and Blood Diseases. In: National Heart Lung and Blood Institute, ed2012
- [Background] Dransfield MT, Bailey WC. COPD: racial disparities in susceptibility, treatment, and outcomes. Clin Chest Med. 2006 Sep;27(3):463-71, vii. doi: 10.1016/j.ccm.2006.04.005. PMID 16880056
- [Background] Akinbami LJ, Liu X. Chronic obstructive pulmonary disease among adults aged 18 and over in the United States, 1998-2009. NCHS Data Brief. 2011 Jun;(63):1-8. PMID 22142836
- [Background] Barr RG, Celli BR, Martinez FJ, Ries AL, Rennard SI, Reilly JJ Jr, Sciurba FC, Thomashow BM, Wise RA. Physician and patient perceptions in COPD: the COPD Resource Network Needs Assessment Survey. Am J Med. 2005 Dec;118(12):1415. doi: 10.1016/j.amjmed.2005.07.059. PMID 16378794
- [Background] Caramori G, Bettoncelli G, Tosatto R, Arpinelli F, Visona G, Invernizzi G, Novelletto BF, Papi A, Adcock IM, Ciaccia A. Underuse of spirometry by general practitioners for the diagnosis of COPD in Italy. Monaldi Arch Chest Dis. 2005 Mar;63(1):6-12. doi: 10.4081/monaldi.2005.651. PMID 16035558
- [Background] Kaminsky DA, Marcy TW, Bachand M, Irvin CG. Knowledge and use of office spirometry for the detection of chronic obstructive pulmonary disease by primary care physicians. Respir Care. 2005 Dec;50(12):1639-48. PMID 16318645
- [Background] Foster JA, Yawn BP, Maziar A, Jenkins T, Rennard SI, Casebeer L. Enhancing COPD management in primary care settings. MedGenMed. 2007 Jul 31;9(3):24. PMID 18092030
- [Background] Stange KC, Zyzanski SJ, Jaen CR, Callahan EJ, Kelly RB, Gillanders WR, Shank JC, Chao J, Medalie JH, Miller WL, Crabtree BF, Flocke SA, Gilchrist VJ, Langa DM, Goodwin MA. Illuminating the 'black box'. A description of 4454 patient visits to 138 family physicians. J Fam Pract. 1998 May;46(5):377-89. PMID 9597995
- [Background] Lusuardi M, De Benedetto F, Paggiaro P, Sanguinetti CM, Brazzola G, Ferri P, Donner CF. A randomized controlled trial on office spirometry in asthma and COPD in standard general practice: data from spirometry in Asthma and COPD: a comparative evaluation Italian study. Chest. 2006 Apr;129(4):844-52. doi: 10.1378/chest.129.4.844. PMID 16608929
- [Background] Walters JA, Hansen EC, Johns DP, Blizzard EL, Walters EH, Wood-Baker R. A mixed methods study to compare models of spirometry delivery in primary care for patients at risk of COPD. Thorax. 2008 May;63(5):408-14. doi: 10.1136/thx.2007.082859. Epub 2007 Nov 16. PMID 18024537
- [Background] Walker PP, Mitchell P, Diamantea F, Warburton CJ, Davies L. Effect of primary-care spirometry on the diagnosis and management of COPD. Eur Respir J. 2006 Nov;28(5):945-52. doi: 10.1183/09031936.06.00019306. Epub 2006 Jul 26. PMID 16870668
- [Derived] Pacheco E, Sohn AJ, Wells C, Sharp LK, Madrid S, Lee TA, Chen YF, Yawn BP, Garcia D, Shim K, Quesada N, Joo MJ. Design of the Reducing Diagnostic Error to Improve Patient Safety (REDEfINE) in COPD and asthma study: A cluster randomized comparative effectiveness trial. Contemp Clin Trials. 2022 Dec;123:106971. doi: 10.1016/j.cct.2022.106971. Epub 2022 Oct 22. PMID 36280032
- See also: Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management and prevention of chronic obstructive pulmonary disease. 2016 — http://www.goldcopd.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met the preliminary eligibility criteria were mailed a recruitment letter with the option to opt out. A phone screen was conducted to confirm eligibility. If eligible, we obtained verbal consent to participate in the study. Their scheduled appointment date was confirmed. They were asked to arrive 90 minutes before their clinic visit for enrollment. Recruitment took place from 07/2017 to 09/2019.
Groups:
- Patient Subject Usual Care: Patients were assigned to the arm group based on the randomization of their primary care provider. The usual care group completed the spirometry test (pre and post BD) during the T4 - 12-month follow-up visit (following the same spirometry protocol as the intervention group did at T0 - baseline visit).
- Patient-Subject Intervention: Patients were assigned to the arm group based on the randomization of their primary care provider. The intervention group completed the spirometry test (pre and post BD) during T0 - baseline visit.
Period: T0: Time of Enrollment - Baseline Visit
Arm/Group | Patient Subject Usual Care | Patient-Subject Intervention
Started | 231 | 171
Completed | 231 | 171
Not Completed | 0 | 0
Period: T1: 3-month Follow-up
Arm/Group | Patient Subject Usual Care | Patient-Subject Intervention
Started | 231 | 171
Completed | 225 | 161
Not Completed | 6 | 10
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 5 | 6
Period: T2: 6-month Follow-up
Arm/Group | Patient Subject Usual Care | Patient-Subject Intervention
Started | 230 | 167
Completed | 225 | 162
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 5
Period: T3: 9-month Follow-up
Arm/Group | Patient Subject Usual Care | Patient-Subject Intervention
Started | 230 | 167
Completed | 225 | 163
Not Completed | 5 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 4 | 4
Period: T4: 12-month Follow-up
Arm/Group | Patient Subject Usual Care | Patient-Subject Intervention
Started | 229 | 167
Completed | 222 | 162
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 7 | 4

BASELINE CHARACTERISTICS:
Population: Intention to treat. Once randomized, patients were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Subject Usual Care | Patient-Subject Intervention | Total
Number analyzed (Participants) | 231 | 171 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (10.4) | 57.5 (10.1) | 57.6 (10.2)
Age, Customized [Count of Participants; unit: Participants]
  40-64 years | 181 | 135 | 316
  65+ years | 50 | 36 | 86
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 119 | 289
  Male | 61 | 52 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 20 | 37
  Not Hispanic or Latino | 214 | 149 | 363
  Unknown or Not Reported | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American/Black | 193 | 139 | 332
  White | 21 | 20 | 41
  Other | 15 | 11 | 26
  Missing | 2 | 1 | 3
Marital Status [Count of Participants; unit: Participants]
  Single/Widowed | 169 | 128 | 297
  Co-habiting/Married | 62 | 43 | 105
Household Income [Count of Participants; unit: Participants]
  < $10,000 | 92 | 71 | 163
  $10,000-19,999 | 41 | 31 | 72
  $20,000-29,999 | 26 | 9 | 35
  $30,000+ | 65 | 51 | 116
  Unknown or Not Reported | 7 | 9 | 16
Education [Count of Participants; unit: Participants]
  High school or less | 107 | 80 | 187
  Vocational/Technical School or Some College | 83 | 61 | 144
  Bachelor and above | 40 | 30 | 70
  Unknown or Not Reported | 1 | 0 | 1
Health Plan [Number; unit: participants]
  Medicaid | 127 | 87 | 214
  Medicare | 60 | 45 | 105
  HMO | 36 | 30 | 66
  PPO | 26 | 21 | 47
  Self-pay | 23 | 13 | 36
  Other | 1 | 0 | 1
Number of Health Plans per Patient [Count of Participants; unit: Participants]
  0-1 | 190 | 146 | 336
  ≥2 | 41 | 25 | 66
Coexisting Conditions [Number; unit: participants]
  Hypertension | 158 | 116 | 274
  Diabetes | 76 | 53 | 129
  Dyslipidemia | 70 | 47 | 117
  Osteoarthritis | 84 | 66 | 150
  Depression | 58 | 37 | 95
  Anxiety | 28 | 23 | 51
  Obstructive/sleep apnea | 21 | 16 | 37
  Congestive Heart Failure | 20 | 9 | 29
  Coronary Artery Disease | 11 | 11 | 22
  Arrhythmia | 21 | 7 | 28
  Autoimmune Disease | 11 | 15 | 26
  Cancer | 12 | 13 | 25
  Osteoporosis | 10 | 7 | 17
  Stroke | 8 | 5 | 13
  End Stage Kidney Disease | 0 | 1 | 1
  Other | 6 | 9 | 15
Number of Coexisting Conditions [Count of Participants; unit: Participants]
  0 | 28 | 16 | 44
  1 | 41 | 29 | 70
  2 | 48 | 47 | 95
  3 | 53 | 37 | 90
  4 | 30 | 23 | 53
  5+ | 31 | 19 | 50
Respiratory Diagnosis [Count of Participants; unit: Participants]
  Asthma | 171 | 127 | 298
  COPD | 28 | 14 | 42
  Asthma and COPD | 32 | 30 | 62
Respiratory Medications [Number; unit: participants]
  Short-acting Bronchodilator | 226 | 169 | 395
  Inhaled Corticosteroids (ICS) | 145 | 107 | 252
  Long-acting muscarinic antagonists (LAMA) | 17 | 11 | 28
  Long-acting beta agonist (LABA) | 2 | 2 | 4
  ICS + LABA | 77 | 60 | 137
  LAMA + LABA | 1 | 1 | 2
Respiratory Symptoms [Number; unit: participants]
  In the past yr., have you had worsened breathing symptoms that caused a change in your medications? | 52 | 29 | 81
  In the past year, have you been hospitalized for breathing problems? | 37 | 14 | 51
  In the past year, have you had the a cough continually for a long time (≥ 3 months)? | 133 | 90 | 223
  In the past year, have you had the a shortness of breath continually for a long time (≥ 3 months)? | 132 | 78 | 210
  In the past year, have you had the a sputum continually for a long time (≥ 3 months)? | 115 | 70 | 185
Number of Respiratory Symptoms [Count of Participants; unit: Participants]
  0 | 62 | 54 | 116
  1 | 42 | 38 | 80
  2 | 43 | 37 | 80
  3 | 84 | 42 | 126
Tobacco Exposure [Count of Participants; unit: Participants]
  Past | 86 | 62 | 148
  Current | 63 | 50 | 113
  Never | 82 | 59 | 141
Second-Hand Smoke Exposure [Count of Participants; unit: Participants]
  Yes | 172 | 132 | 304
  No | 59 | 39 | 98
Illicit Substance Use [Number; unit: participants]
  Yes | 26 | 26 | 52
  Would rather not say | 1 | 0 | 1
Modified Medical Research Council Dyspnea Scale [Count of Participants; unit: Participants]
  0 = only breathless with strenuous exercise | 49 | 35 | 84
  1 = short of breath when hurrying or walking up a slight hill | 73 | 60 | 133
  2 = walk slower or have to stop for breath when walking | 48 | 34 | 82
  3 = stop for breath after walking about 100 yards or a few minutes | 50 | 34 | 84
  4 = too breathless to leave the house or when dressing | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Healthcare Visits
Description: Determine differences in healthcare visits which include all-cause and respiratory related, acute care outpatient visits, emergency department visits, and hospitalizations between groups
Time Frame: 1 year
Population: Intention to treat. Once randomized, patients were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Subject Usual Care | Patient-Subject Intervention
Number analyzed (Participants) | 231 | 171
Participants
  Emergency room visit: Yes | 111 | 76
  Emergency room visit: No | 119 | 93
  Emergency room visit: Missing | 1 | 2
  Hospitalization: Yes | 48 | 17
  Hospitalization: No | 182 | 152
  Hospitalization: Missing | 1 | 2
  Acute outpatient visit: Yes | 61 | 35
  Acute outpatient visit: No | 169 | 134
  Acute outpatient visit: Missing | 1 | 2
  Routine primary care visits: Yes | 198 | 138
  Routine primary care visits: No | 32 | 31
  Routine primary care visits: Missing | 1 | 2
  New diagnostic tests: Yes | 126 | 72
  New diagnostic tests: No | 104 | 97
  New diagnostic tests: Missing | 1 | 2

2. Secondary Outcome: Total With Diagnosis of COPD and/or Asthma Consistent With Spirometry Results
Description: determine differences in the accuracy of diagnosis between groups
Time Frame: 1 year
Population: This analysis was only done for patients who had clear yes or no diagnosis accuracy from spirometry. This also excluded those did not have missing spirometry either due to withdraw or lost to follow-up. Two patients with yes or no diagnosis accuracy from spirometry withdrew, but they were either qualified for "Correct initial diagnosis" or "Ever remove wrong initial diagnosis" and thus lead to no missing in this table.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Subject Usual Care | Patient-Subject Intervention
Number analyzed (Participants) | 176 | 128
Participants
  Correct initial diagnosis | 76 | 55
  Stayed with wrong initial diagnosis | 92 | 64
  Ever removed wrong initial diagnosis | 8 | 9

ADVERSE EVENTS:
Time Frame: T0-T4. From the enrollment time until the end of the 12-month follow-up visit.
Arm/Group | Patient Subject Usual Care | Patient-Subject Intervention
All-Cause Mortality (participants affected / at risk) | 1/231 | 0/171
Serious Adverse Events (participants affected / at risk) | 0/231 | 0/171
Other Adverse Events (participants affected / at risk) | 0/231 | 0/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT03137303/Prot_SAP_000.pdf